CLINICAL TRIAL: NCT06054113
Title: An Open-label, Multicenter, Phase 2 Study to Evaluate Efficacy, Safety, and Pharmacokinetics (PK) of Blinatumomab in Chinese Pediatric Subjects With Relapsed or Refractory B Precursor Acute Lymphoblastic Leukemia (R/R B-ALL)
Brief Title: Study of Blinatumomab Administration in Chinese Pediatric Participants With Relapsed/Refractory B Precursor Acute Lymphoblastic Leukemia (R/R B-ALL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190359
Record Dates: First submitted 2023-09-18; First posted 2023-09-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: B Precursor Acute Lymphoblastic Leukemia; Relapsed/Refractory B Precursor Acute Lymphoblastic Leukemia
Keywords: Relapsed/Refractory B precursor Acute Lymphoblastic Leukemia; R/R B-ALL; Blinatumomab
MeSH Terms: conditions — Recurrence | interventions — blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Blinatumomab (Experimental): Participants will receive up to 5 cycles of blinatumomab (cycle is 42 days), including a 28-day continuous intravenous infusion (CIVI) of blinatumomab and a 14-day treatment free interval.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Administered via CIVI
  Other Names: Blincyto®

SUMMARY:
The primary objective of this study is to evaluate the efficacy of blinatumomab.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent or legally authorized representative has provided informed consent when the participant is legally too young to provide informed consent and the participant has provided written assent based on local regulations and/or guidelines prior to any study-specific activities/procedures being initiated
* Pediatric participants aged > 1 month and < 18 years at the time of informed consent
* Relapsed or/refractory precursor B-cell acute lymphoblastic leukemia (ALL) disease, defined as ≥5% bone marrow blasts with at least one of the following:
* Second or later bone marrow relapse;
* Any marrow relapse after allogeneic hematopoietic stem cell transplant (alloHSCT);
* Refractory to other treatments:
* For participants in first relapse: failure to achieve a complete remission (CR) following a full standard reinduction chemotherapy regimen
* For participants who have not achieved a first remission, failure to achieve remission following a full standard induction regimen
* Karnofsky performance status ≥ 50% for participants ≥ 16 years
* Lansky performance status ≥ 50% for participants < 16 years

Exclusion Criteria:

- Evidence of current central nervous system (CNS) involvement by ALL. Participants with CNS disease at the time of relapse are eligible if CNS is successfully treated prior to enrollment.

Other Medical Conditions

* Clinically relevant CNS pathology requiring treatment (eg, unstable epilepsy).
* Isolated extramedullary (EM) disease.
* Active malignancy other than ALL.
* Burkitt's leukemia according to the World Health Organization (WHO) 2016 criteria.
* Abnormal renal or hepatic function at screening as defined below:
* Abnormal serum creatinine based on age/gender as described by Threshold Creatinine Values
* Direct bilirubin > 1.5 mg/dl (25.6 μmol/L) at screening (unless related to Gilbert's or Meulengracht disease).
* Symptoms and/or clinical signs and/or radiological and/or sonographic signs that indicate an acute or uncontrolled chronic infection, any other concurrent disease or medical condition that could be exacerbated by the treatment or would seriously complicate compliance with the protocol.
* Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (hepatitis B surface antigen [HBsAg] positive) or hepatitis C virus (HCV) (anti-HCV positive).
* Known hypersensitivity to blinatumomab or any of the products or components of the blinatumomab formulation.

Prior/Concomitant Therapy

* AlloHSCT within 12 weeks prior to start of protocol-specified therapy.
* Active acute or chronic Graft-versus-Host-Disease (GvHD) requiring systemic treatment with immunosuppressive medication.
* Radiotherapy within 2 weeks prior to start of protocol-specified therapy.
* Immunotherapy (eg, rituximab) within 4 weeks prior to start of protocol-specified therapy. Prior failed cluster of differentiation 19 (CD19) directed therapy such as prior blinatumomab or CD19 chimeric antigen receptor T cells (CAR T cell) will be allowed (with demonstrated continued CD19+ expression) if treatment ended > 4 weeks prior to start of protocol-specified therapy.
* Cancer chemotherapy within 2 weeks before the start of protocol-specified therapy. With the exception of intrathecal chemotherapy and/or low dose maintenance therapy for example vinca alkaloids, mercaptopurine, methotrexate, or hydroxyurea or pre-phase chemotherapy and/or dexamethasone. Any low dose chemotherapy as stated above must be discontinued before starting pre-phase.

Prior/Concurrent Clinical Study Experience

- Currently receiving treatment in another investigational device or drug study, or less than 4 weeks since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.

Other Exclusions

* Female participants of childbearing potential with a positive pregnancy test assessed at Screening by a highly sensitive urine or serum pregnancy test.
* Female participants who are breastfeeding or who plan to breastfeed while on study through 12 months after the last dose of protocol-required treatment with highest teratogenic risk.
* Female participants of childbearing potential unwilling to use protocol-specified method of contraception during treatment and for an additional 12 months after the last dose of protocol-required treatment with highest teratogenic risk.
* Male participants with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use contraception during treatment and for an additional 6 months after the last dose of protocol-required therapy with highest teratogenic risk.
* Participant likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participant and investigator's knowledge.
* Female participants planning to become pregnant while on study through 12 months after the last dose of protocol-required treatment with highest teratogenic risk.
* Male participants unwilling to abstain from donating sperm during treatment and for an additional 6 months after the last dose of protocol-required treatment with highest teratogenic risk.

Ages: 1 Month to 204 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2027-10-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Complete Remission (CR) | Up to 84 days
Number of Participants with CR with Partial Recovery of Peripheral Blood Counts (CRh) | Up to 84 days

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 240 days
Number of Participants with Serious TEAEs | Up to approximately 2 years
Number of Participants with Treatment-related TEAEs | Up to approximately 240 days
Number of Participants with Adverse Events of Interest | Up to approximately 240 days
Steady State Concentration (Css) of Blinatumomab | Days 3, 8, 9 and 29
Clearance of Blinatumomab | Days 3, 8, 9 and 29
Overall Survival (OS) Rate | Up to approximately 2 years
Relapse-Free Survival (RFS) Rate | Up to approximately 2 years
Number of Participants who Receive Allogeneic Hematopoietic Stem Cell Transplant (alloHSCT) | Up to approximately 2 years
100-day Mortality Rate After alloHSCT | Up to approximately 2 years
Number of Participants with Anti-blinatumomab Antibody (ADA) Formation | Up to approximately 240 days
Minimal Residual Disease (MRD) Response | Up to 84 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- China (7):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Childrens Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Wuhan Childrens Hospital, Wuhan, Hubei
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com